CLINICAL TRIAL: NCT02775799
Title: Prospective Multi-center National Swiss Sarcoma Cohort Study
Brief Title: National Swiss Sarcoma Cohort Study
Acronym: SwissSARCOS
Status: Terminated | Type: Observational
Why Stopped: Principal Investigator has left the Institution
Sponsor: Balgrist University Hospital (Other)
Collaborators: University of Bern (Other)
Responsible Party: Sponsor
Other Study IDs: 2014-0394
Record Dates: First submitted 2016-05-16; First posted 2016-05-18 (Estimated); Last update posted 2018-10-02 (Actual); Status verified 2018-09

CONDITIONS: Sarcoma; Neoplasm of Bone; Neoplasms; Soft Tissue Sarcoma; Soft Tissue Neoplasm; Sarcoma of Bone
MeSH Terms: conditions — Sarcoma; Bone Neoplasms; Neoplasms; Soft Tissue Neoplasms; Osteosarcoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Registration — Registration according to approved data sets

SUMMARY:
Registration of all sarcoma patients treated at a specialized sarcoma center in Switzerland.

DETAILED DESCRIPTION:
SCIENTIFIC BACKGROUND OF STUDY, EXPECTED OUTCOME, AND RELEVANCE Sarcomas represent malignant bone and soft tissue tumours. Overall, these are very rare tumours representing less than 1% of all cancers (besides carcinomas and haematological cancers). Furthermore, with the advent of molecular knowledge, more than 100 subtypes of sarcomas can be distinguished and many of them share a distinct biological behaviour opening the possibility of targeted therapy. The management of patients with sarcomas is extremely complex and highly multidisciplinary, involving the pathologist, the orthopaedic oncologist, a paediatric and medical oncologist, the radiation oncologist, the reconstructive as well as visceral and chest surgeon. Surgery remains the mainstay of treatment, but almost always in combination with either radiotherapy or chemotherapy, or novel targeted therapy. The key of successful therapy (and consequent successful outcome for the patient) remains the orchestrated team approach among these disciplines where the therapeutic strategy is interdisciplinary determined at the sarcoma board. Unfortunately, all too often and still nowadays, patients also in Switzerland are not treated within such a network. E.g., too many surgeons still believe that they are capable to remove a soft tissue lump (which technically is true), just to send the patient off after surgery to the medical oncologist, and never see the patient again. All too often this may result for example in an unnecessary amputation, a devastating consequence for the patient. A surgeon needs to be aware of the interpretation of the pathologic specimen, the possibilities of adjuvant treatment, and most importantly, the biology of each subtype of sarcoma, before embarking on surgery. Because of all the reasons listed above, it is very reasonable to centralize the treatment of sarcoma patients to improve the treatment and outcome for sarcoma patients in Switzerland, as is foreseen by the current initiative of HSM by the GDK. It is very important to state that such uncoordinated treatment of sarcoma patients with the potential deleterious consequences is an international phenomenon. Many groups have independently established that the lack of interdisciplinarity leads to worse patient outcome and survival. Many reasons account for this: rarity of disease, lack of knowledge, lack of awareness, and all too often also pride and prestige. The only way out is to bring treating physicians together and to make the institutions aware that applying simple management strategies -such as coordinated treatment- does improve the outcome of sarcoma patients, which has been proven in many countries already. Nowadays in Switzerland, there are only very few groups/institutions who deal exclusively with sarcoma patients. Consequently, the therapeutic approach and quality are varying a lot. Therefore, the establishment of a Swiss Sarcoma Cohort Study (SwissSARCOS) is instrumental in improving the quality of treatment, which has already been shown in other countries. If all patients are registered including their respective follow-up, the type of treatment can be registered and the various geographic regions can be compared with respect to patients' outcome. It can be expected that the awareness of treating a sarcoma patient according to international standards will be increased, for the benefit of the patient. Importantly, such registration will provide the base to participate in international studies in form of clinical trials, which is a prerequisite and also requested by the HSM, and will further improve the quality of the therapy of sarcoma patients in Switzerland. Such cohort study will also allow to assess the prevalence of sarcoma types in Switzerland, with its associated regional differences. Because of its rarity, registering all sarcoma types in Switzerland will bring together sizeable numbers and therefore will provide the base for numerous outcome studies. Because it is known that sarcomas are extremely heterogeneous and are molecularly defined, studying molecular alterations in tumour tissue is essential to advance the field. The French Sarcoma Group (Prof. JM.Coindre, F.Chibon) has started such initiative decades ago and are therefore leaders in this field. The investigators therefore speculate that SwissSARCOS ultimately will also provide a strong base to establish a sarcoma tissue bank which allows the study of molecular alterations on the one hand, but on the other hand to correlate these findings with clinical outcome. For these reasons outlined above, the establishment of SwissSARCOS is crucial to improve treatment quality of sarcoma patients in Switzerland.

The specific questions addressed within the first 2-year time period include: 1.) what is the prevalence of which sarcoma type in Switzerland; 2.) What is the quality of the (correct) diagnosis?; 3.) What is the quality of treatment?; 4.) What is the outcome (survival, local recurrence, metastasis etc.) of sarcoma patients in Switzerland? Complete identification and thorough assessment of the basic clinical parameters ("minimal data set") of sarcoma patients treated in Switzerland in a prospective manner will allow to improve the quality of patient care as outlined above. This is also in line with the national strategy to register all cancer patients. Therefore, this effort is very timely and has direct impact on public health issues. As shown for other cohort studies in Switzerland (e.g. HIV), such assessment of clinical parameters has widespread implications not only on the standard of patient care, but also on addressing important clinical research questions, thereby becoming a very relevant health care issue. Through such coordinated and orchestrated approach, Switzerland will become a key player for international collaborations to improve the treatment for sarcoma patients. It is very clear that it cannot be expected to include every single patient diagnosed with sarcoma of whole Switzerland right from the beginning. Obviously, it is the intention to first set a strong base with national key players and institutions, and then to strengthen this collaborative network to become a national instrument. The network of national key players and institutions should allow to bring all the regional efforts to a national level. The Sarcoma Center Zurich (www.sarkomzentrum.ch) is certified as a center of excellence by the German Cancer Society (DKG= Deutsche Krebsgesellschaft) since December 2013, the very first one in Switzerland. The Sarcoma Center in Zurich bases on the instrumental efforts of the cantonal government ("Regierungsrat") to specifically support the multidisciplinary team approach in musculoskeletal oncology, both on the clinical and research side since 2010 by the HSM program (www.sarkomboard.ch). Over the years, collaboration with all major regional hospitals in Switzerland was set up. All the collaborators of these hospitals have assembled to strengthen the goal to build up a Sarcoma Cohort Study. For that reasons the Sarcoma Center Zurich has the lead for this multicentre study and the ethic committee of Zurich is chosen as the leading committee.

Future: Molecular analyses of sarcoma tissue are the key for the advancement of the treatment strategies of sarcoma patients. Again based on the HSM program funded by the cantonal government in Zurich, tumour tissue specimens as well as blood is collected and stored of each single patient operated for a sarcoma in Zurich. This allows addressing fundamental molecular questions via TMA (tissue microarray analyses), the characterization of molecular markers, both in-vitro and in-vivo, proteomic diagnostic analyses, and novel targeted treatment approaches (please refer to www.sarkomzentrum.ch). It is foreseen that in the second phase of this grant project -and after having established the fundamentals of the national cohort study- to extend the efforts to not only gather patient data ("minimal data set"), but also tumour tissue/blood from the sarcoma patients treated in Switzerland.

In a further next step, and again based on these efforts outlined above with a nationally well documented patient cohort, the base will be set to participate in international clinical trials to test for example novel drug compounds or novel diagnostic imaging tools.

ELIGIBILITY:
Inclusion Criteria:

* all primary bone and soft tissue sarcoma defined by th WHO classification 2013

Exclusion Criteria:

* all non- primary sarcomas
* patient's wish

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients diagnosed with histo- pathological proven sarcoma
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2015-04; Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Overall survival rate | up to 20 years after first line treatment

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Fuchs, MD PhD, Study Chair — Balgrist UH
Locations (1):
- Balgrist University Hospital, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Assessed data shall be shared with the National Institute for Cancer Epidemiology an Registration and the cantonal cancer registers